CLINICAL TRIAL: NCT04427826
Title: Efficacy of Morphine in Reducing the Rate of Early Non-Invasive Ventilation (NIV) Failure in Acute Exacerbation of Chronic Obstructive Pulmonary Disease (COPD), Phase I/IIa
Brief Title: Efficacy of Morphine in Reducing the Rate of Early Non-Invasive Ventilation Failure in Acute Exacerbation of Chronic Obstructive Pulmonary Disease, Phase I/IIa
Acronym: MORPHEUS I/IIa
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-004274-25; 2019-004274-25 (EudraCT Number)
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Acute exacerbation; COPD; NIV; Morphine; DLT
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Phase I / IIa prospective, monocentric and open therapeutic study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient admitted for acute Exacerbation of Chronic Obstructive (Experimental): Patient admitted for acute Exacerbation of Chronic Obstructive Pulmonary Disease (COPD) and required NIV
  Interventions: Drug: Morphine hydrochloride

INTERVENTIONS:
Drug: Morphine hydrochloride — A single open-label injection of morphine (T0) at the dose closest to that defined by the model (estimation by Bayesian method) from among the following 4 doses: 0.02; 0.04; 0.07 and 0.1mg/kg will be adminestred to the patients.

SUMMARY:
Acute exacerbations of Chronic Obstructive Pulmonary Disease (COPD) are a major source of morbidity and mortality for patients and cost to the society. In case of acute respiratory failure with hypercapnia and acidosis, Non Invasive Ventilation (NIV) is preferred as a first line treatment.

NIV failures are not uncommon, from 15% in intensive care to 25 - 30% in emergency departments. They most often occur at the start of the NIV or in the hours that follow. There are many reasons for these failure. Among these are; dyspnea, discomfort, the pain related to the exacerbation and also to the NIV are frequently noted.

The use of certain drugs with anxiolytic, hypnotic and/or analgesic properties could also be useful. Some sedatives and opioids have already been studied in this indication but without a therapeutic trial and satisfactory methodology. Among the molecules of interest, Morphine seems interesting . It's administration could reduce the ventilatory rate, intensity of dyspnea, pain and anxiety as well as dynamic hyperinflation.

The investigators believe that morphine administration will decrease the rate of early NIV failure by improving comfort (decreased dyspnea and pain) and ventilation (decreased respiratory rate and increase in tidal volume) in patients with exacerbations of COPD.

However, before considering a randomized phase III efficacy study, it is necessary to determine the optimal dose of morphine in this indication, through a phase I/II dose-finding study taking into accounts both the efficacy and toxicity of morphine.

The main objective of this study, is to determine the optimal dose of morphine administered at the initiation of NIV in patient with acute Exacerbation of Chronic Obstructive Pulmonary Disease (COPD), which is defined as the maximum gain function combining the probability of dose-limiting toxicity with PaCO2.Therefore, the impact of morphine administration on the physiological parameters of NIV- COPD exacerbation patients will be assessed.

DETAILED DESCRIPTION:
Patients included in this dose-finding study will be enrolled consecutively after consent and verification of the selection criteria, with a minimum of 24 hours after completion of previous patient follow-up.

Prior to the administration of morphine, the following exams will be performed: clinical, paraclinical and biological parameters.

NIV will be started and performed in BiPAP pressure mode with facial mask. A Tidal Volume (Vt) to the maximum of 6 - 8ml/kg, an expiratory positive airway pressure (EPAP) of 5cm H2O and the FiO2 set at 35%. The settings will be adapted according to the SpO2 (88%≤SpO2≤92%) and the clinical tolerance.

Thereafter, the patients included will receive a single open-label injection of morphine (T0) at the dose closest to that defined by the model (estimation by Bayesian method) from among the following 4 doses: 0.02; 0.04; 0.07 and 0.1mg/kg.

A double check of the preparation of the dose administered will be carried out by a physician and a nurse in an emergency department.

Each result is aimed to refine the gain function which will be used to estimate the optimal dose for the next patient. The dose to be administered to the next patient will be determined by the Clinical Investigation Centre based on the data of the previous patient. It will be determined using a gain function whose objective is to represent the best compromise between efficacy and safety. It assigns a value to the patient representing the benefit: in case of toxicity this value will be 0; otherwise it will be equal to the decrease in PaCO2.

Constant monitoring for up to 4 hours will be done as part of this study to detect the occurrence of adverse events. In particular, the following will be monitored: disturbances of consciousness, vomiting or secretions requiring airway protection; hemodynamic instability; restlessness and/or inability to keep the mask on. Therefore, ongoing monitoring for routine patient care may be extended at the discretion of the clinical physician in charge of the patient.

Follow-up of patients will be done in 15 minutes, 1 hour, 4 hours (or NIV stop) and 24 hours. Clinical, paraclinical, biological parameters and the occurrence of adverse events will be performed in 15 minutes, 1 and 4 hours follow-up. During 24 hours only the occurrence of adverse event will be reported.

The trial shall be concluded when the maximum number of patients is reached (N=24), or when a sufficiently accurate estimate of the dose maximizing the benefit-risk balance is obtained while remaining within the toxicity limit set at a 30% probability of DLT. The precision of this estimate will be measured by the ratio of the upper and lower bounds of the confidence interval. If this ratio is less than 5, the precision is considered to be sufficient to stop the study.

Four groups of data will be collected at different times: biological parameter, clinical and paraclinical parameters as well adverse event.

Clinical parameter: demographic variable (gender, age), weight, height, BMI, Richmond Agitation- Sedation Scale, Visual analog scale of dyspnea (Borg scale), numerical rating scale for pain assessment.

Paraclinical parameter: Vital parameters: heart rate, respiratory rate, blood pressure, ventilatory rate, SpO2, NIV settings, EPAP, IPAP and Tidal Volume.

Biological parameter: Blood count, arterial blood gas, chemistry panel.

outcome measure: Optimal dose is defined as the dose associated with the maximum of gain function, used to determine the best compromise between efficacy and toxicity.

It combines:

1. The probability of dose - limiting toxicity (DTL), defined as the occurrence of one or more of the following criteria occurring within 4 hours of morphine administration:

   * Respiratory Rate ≤ 10/min;
   * Richmond Agitation-Sedation Scale (RASS) < -2
   * Vomiting
   * Naloxone administration.
2. Efficacy and toxicity defined by:

   * PaCO2 1 hour after morphine injection, according to the hormetic dose-response model ("J-curve": efficacy first increases with the dose, then reach a maximum and decreases in case of excessive bradypnea).

Study design:

Estimation of enrollment: Up to 24 participants. The calculation of the sample size was carried out by simulating several scenarios based on the prior to be used in the study. The simulated scenarios are as follows: one with low toxicity (5% at 0.02 mg/kg and 30% at 0.1 mg/kg), one with high toxicity (10% at 0.02 mg/kg and 40% at 0.04 mg/kg) and one where the toxicity is identical to the prior.

Simulation results showed a number of subjects required up to 24, with a median of 6 to 11, according to the scenario. The investigators therefore chose to define a maximum number of patients to 24, which is higher than the average of the worst-case scenario and corresponds to the maximum number of patients required among the 100 simulations of the worst-case scenario. However, it is very likely that the inclusions will be stopped earlier, when the accuracy is satisfactory.

Analysis:

The method used will be an adaptive Bayesian dose-finding procedure for a binary response (DLT), and a continuous response (PaCO2 used as a biomarker of efficacy and toxicity, following a hormetic response), using a gain function which objectively represent the compromise between efficiency and safety. The investigators will use a function already described in the literature .

No interim analysis planned for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients Aged ≥ 18 years
* Current or former smoker at least 10 packs-years
* Patient with a history of COPD according to the Gold guidelines , after review of the medical record by the physician in charge
* Acute exacerbation of COPD (greater degradation of respiratory symptoms than the usual daily variations and requiring a modification of therapeutic management)
* Need to implement NIV treatment (respiratory acidosis with pH<7.35)
* Ventilation frequency > 20min
* Affiliation to the French security system (or equivalent)
* Written informed consent from the patient or his surrogates. In patients who are not able to consent on admission an emergency inclusion procedure will be allowed, with a mandatory delayed consent.

Exclusion Criteria:

* Patient already treated by NIV during admission (e. g. introduction in pre-hospital by SMUR) or started more than one hour ago in the department.
* Sedative (barbiturates, benzodiazepines and related substances and other sedatives) or morphine treatment within 24 hours before inclusion
* Chronic alcoholism
* Contra-indication to NIV: disturbances of consciousness (Glasgow < 11) except moderate hypercapnic encephalopathy; indication of immediate intubation; risk of inhalation; sputum impossible; hemodynamic instability; inability to remove the mask; trauma, surgery or facial malformation; patients with pH < 7.25 can only be included in intensive care unit or in the vital emergency room of the emergency department, under continuous monitoring
* NIV with palliative purpose from the outset with death expected within 24 hours of inclusion
* Non-communicative patient or significant dementia making them unable to participate in the study
* Contra-indication to morphine without acute respiratory distress
* Pregnant or breastfeeding women
* Major mentioned in Articles L1121-6 and 1121-8 of French public health cod
* Patients in a period of exclusion from other research involving the human person type 1 or 2
* Subject cannot be contacted in case of emergency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
The probability of dose - limiting toxicity (DTL), defined as the occurrence of one or more of the following criteria occurring within 4 hours of morphine administration | 4 hours
  Respiratory Rate ≤ 10/min; Richmond Agitation-Sedation Scale (RASS) < -2;Vomiting and Naloxone administration
Efficacy and toxicity | 1 hour
  PaCO2 1 hour after morphine injection, according to the hormetic dose-response model

SECONDARY OUTCOMES:
Percentage of adverse events | 1, 4 and 24 hours
  Percentage of adverse event occurred

CONTACTS AND LOCATIONS:
Overall Officials: Damien VIGLINO, MD, PhD, Principal Investigator — Grenoble Alpes University Hospital, HP2 laboratory - INSERM U1042 and Grenoble Alpes University
Locations (1):
- Emergency Department of Grenoble Alpes University Hospital, Grenoble, Isère, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: Yes
The international writing and publication rules (The Uniform Requirements for Manuscripts of the ICMJE, April 2010) will be followed. The minimum anonymized source data for performing the statistical analysis will be made public at the time of publication, with the article, or deposited in an appropriate public database. Other anonymized data may be available from the principal investigator upon reasonable request and with the consent of the sponsor.
  In accordance with the French law n ° 2002-303 of March 4th, 2002, the subjects can be informed, at their request, of the overall results of the research. In this study, the investigators commit to individually communicating the overall results to each subject participating in the research by a short (popularized) summary and associated with a copy of the scientific article.
Supporting Information: Study Protocol, SAP
Time Frame: At the time of publication
Access Criteria: The international writing and publication rules (The Uniform Requirements for Manuscripts of the ICMJE, April 2010) will be followed. And In accordance with the French law n ° 2002-303 of March 4th, 2002

REFERENCES:
- [Background] Wedzicha JA Ers Co-Chair, Miravitlles M, Hurst JR, Calverley PM, Albert RK, Anzueto A, Criner GJ, Papi A, Rabe KF, Rigau D, Sliwinski P, Tonia T, Vestbo J, Wilson KC, Krishnan JA Ats Co-Chair. Management of COPD exacerbations: a European Respiratory Society/American Thoracic Society guideline. Eur Respir J. 2017 Mar 15;49(3):1600791. doi: 10.1183/13993003.00791-2016. Print 2017 Mar. PMID 28298398
- [Background] Bounes V, Charriton-Dadone B, Levraut J, Delangue C, Carpentier F, Mary-Chalon S, Houze-Cerfon V, Sommet A, Houze-Cerfon CH, Ganetsky M. Predicting morphine related side effects in the ED: An international cohort study. Am J Emerg Med. 2017 Apr;35(4):531-535. doi: 10.1016/j.ajem.2016.11.053. Epub 2016 Nov 30. PMID 28117179
- [Result] Vogelmeier CF, Criner GJ, Martinez FJ, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Chen R, Decramer M, Fabbri LM, Frith P, Halpin DM, Lopez Varela MV, Nishimura M, Roche N, Rodriguez-Roisin R, Sin DD, Singh D, Stockley R, Vestbo J, Wedzicha JA, Agusti A. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report. GOLD Executive Summary. Am J Respir Crit Care Med. 2017 Mar 1;195(5):557-582. doi: 10.1164/rccm.201701-0218PP. PMID 28128970
- [Result] Halbert RJ, Natoli JL, Gano A, Badamgarav E, Buist AS, Mannino DM. Global burden of COPD: systematic review and meta-analysis. Eur Respir J. 2006 Sep;28(3):523-32. doi: 10.1183/09031936.06.00124605. Epub 2006 Apr 12. PMID 16611654
- [Result] Schmidt SA, Johansen MB, Olsen M, Xu X, Parker JM, Molfino NA, Lash TL, Sorensen HT, Christiansen CF. The impact of exacerbation frequency on mortality following acute exacerbations of COPD: a registry-based cohort study. BMJ Open. 2014 Dec 19;4(12):e006720. doi: 10.1136/bmjopen-2014-006720. PMID 25526796
- [Result] Hartl S, Lopez-Campos JL, Pozo-Rodriguez F, Castro-Acosta A, Studnicka M, Kaiser B, Roberts CM. Risk of death and readmission of hospital-admitted COPD exacerbations: European COPD Audit. Eur Respir J. 2016 Jan;47(1):113-21. doi: 10.1183/13993003.01391-2014. Epub 2015 Oct 22. PMID 26493806
- [Result] Mackay AJ, Hurst JR. COPD exacerbations: causes, prevention, and treatment. Med Clin North Am. 2012 Jul;96(4):789-809. doi: 10.1016/j.mcna.2012.02.008. Epub 2012 Mar 16. PMID 22793945
- [Result] Rochwerg B, Brochard L, Elliott MW, Hess D, Hill NS, Nava S, Navalesi P Members Of The Steering Committee, Antonelli M, Brozek J, Conti G, Ferrer M, Guntupalli K, Jaber S, Keenan S, Mancebo J, Mehta S, Raoof S Members Of The Task Force. Official ERS/ATS clinical practice guidelines: noninvasive ventilation for acute respiratory failure. Eur Respir J. 2017 Aug 31;50(2):1602426. doi: 10.1183/13993003.02426-2016. Print 2017 Aug. PMID 28860265
- [Result] Osadnik CR, Tee VS, Carson-Chahhoud KV, Picot J, Wedzicha JA, Smith BJ. Non-invasive ventilation for the management of acute hypercapnic respiratory failure due to exacerbation of chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2017 Jul 13;7(7):CD004104. doi: 10.1002/14651858.CD004104.pub4. PMID 28702957
- [Result] Ko BS, Ahn S, Lim KS, Kim WY, Lee YS, Lee JH. Early failure of noninvasive ventilation in chronic obstructive pulmonary disease with acute hypercapnic respiratory failure. Intern Emerg Med. 2015 Oct;10(7):855-60. doi: 10.1007/s11739-015-1293-6. Epub 2015 Sep 4. PMID 26341216
- [Result] Maignan M, Chauny JM, Daoust R, Duc L, Mabiala-Makele P, Collomb-Muret R, Roustit M, Maindet C, Pepin JL, Viglino D. Pain during exacerbation of chronic obstructive pulmonary disease: A prospective cohort study. PLoS One. 2019 May 24;14(5):e0217370. doi: 10.1371/journal.pone.0217370. eCollection 2019. PMID 31125359
- [Result] Yeung WY, Reigner B, Beyer U, Diack C, Sabanes Bove D, Palermo G, Jaki T. Bayesian adaptive dose-escalation designs for simultaneously estimating the optimal and maximum safe dose based on safety and efficacy. Pharm Stat. 2017 Nov;16(6):396-413. doi: 10.1002/pst.1818. Epub 2017 Jul 9. PMID 28691311
- [Result] Jolliet P, Ouanes-Besbes L, Abroug F, Ben Khelil J, Besbes M, Garnero A, Arnal JM, Daviaud F, Chiche JD, Lortat-Jacob B, Diehl JL, Lerolle N, Mercat A, Razazi K, Brun-Buisson C, Durand-Zaleski I, Texereau J, Brochard L; E.C.H.O. ICU Trial Investigators. A Multicenter Randomized Trial Assessing the Efficacy of Helium/Oxygen in Severe Exacerbations of Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2017 Apr 1;195(7):871-880. doi: 10.1164/rccm.201601-0083OC. PMID 27736154
- [Result] Lightowler JV, Wedzicha JA, Elliott MW, Ram FS. Non-invasive positive pressure ventilation to treat respiratory failure resulting from exacerbations of chronic obstructive pulmonary disease: Cochrane systematic review and meta-analysis. BMJ. 2003 Jan 25;326(7382):185. doi: 10.1136/bmj.326.7382.185. PMID 12543832